CLINICAL TRIAL: NCT03524443
Title: Evaluation of Art-therapy on Alexithymia in Patients Suffering From Anorexia Nervosa and From Bulimia,a Pilot Study
Brief Title: Evaluation of Art-therapy on Alexithymia in Patients Suffering From Anorexia Nervosa and From Bulimia
Acronym: ALEXART
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0180; 2018-A01285-50 (Other: ID-RCB)
Record Dates: First submitted 2018-05-02; First posted 2018-05-14 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Anorexia Nervosa/Bulimia
Keywords: Affective symptom; Art Therapy; alexithymia; emotional disturbance; hyperphagia; psychotherapy; rehabilitation; factor of resistance
MeSH Terms: conditions — Anorexia Nervosa; Bulimia; Affective Symptoms; Hyperphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient suffering from anorexia/bulimia: Each patient will receive standard care: multidisciplinary and corresponding to the HAS recommendations for anorexia nervosa and bulimia nervosa associated with semimonthly or weeklies sessions of art therapy treatment, using all types of art, realized by trained professional, in Toulouse. Each patient will be her own control before art therapy Female patients with anorexia nervosa or bulimia according to DSM-5 criteria, patient will be above 16 years-old
  Interventions: Behavioral: Art Therapy treatment

INTERVENTIONS:
Behavioral: Art Therapy treatment — The main objective is to describe the evolution at 3 months on the alexithymic dimension in the course of a treatment in art therapy, in patients with anorexia nervosa or bulimia.
  Art therapy is a generic term grouping different artistic disciplines adapted and used for therapeutic purposes. It is through commitment to creative work that the therapeutic work of elaboration and reflection takes place in contrast to verbal psychotherapies and mediated psychotherapies that use speech as the main therapeutic tool. All forms of practice referring to categories of art can be used: painting, music, modeling, dance, theater and writing

SUMMARY:
Alexithymia is often found in patients suffering from anorexia nervosa or from bulimia. Art-therapy is widely used in this indication without there is a study in the literature assessing it. ALEXART is an observational prospective multicenter cohort pilot study, assessing the effect at 3 months of art therapy on alexithymia, in patients presenting anorexia nervosa or bulimia.

DETAILED DESCRIPTION:
Alexithymia, defined by difficulties to identify and describe feelings as well as a poverty of imaginary life, is found in patients with anorexia nervosa (AN) or bulimia (BN) in numerous studies. Some publications show that it is a factor of resistance in several forms of psychotherapies and of poor prognosis for these patients who already present a high rate of chronification and mortality because of the complications of the undernutrition and the suicide risk. Art therapy is very wide-spread in the care of AN and of BN, but little studied. About alexithymia, if there is no psychotherapy having made the proof of its efficiency currently, some studies suggest the interest of art-therapy on alexithymic features, but none, to our knowledge, estimated the effect.

The investigator suggest to describe the evolution at 3 months of art therapy on alexithymia, using the Toronto Alexithymia Scale in 20 items (TAS-20), in patients with AN or BN. The investigators shall also describe the evolution at 3 months with the TAS-20 as well as the relationship between variations of alexithymia and BMI in patients presenting AN at 1 and 3 months globally and in each of the centers. The investigators will also evaluate the effect of depression and anxiety at 1 and 3 months of art therapy on alexithymia.The investigators shall realize an observational prospective multicenter cohort study design. Each patient will receive standard care: multidisciplinary and corresponding to the HAS recommendations and semimonthly or weeklies sessions of art therapy, using all types of art. Thus, each patient will be her own control before art therapy.

ELIGIBILITY:
Inclusion Criteria:

* to be a woman, aged 16 or more, having DSM-5 diagnosis of anorexia nervosa or bulimia nervosa, inpatient in "Psychiatry, Psychotherapy and Art Therapy" ward at CHU de Toulouse or at " clinique Castelviel " in Toulouse.

Exclusion Criteria:

* acute psychotic symptoms
* pregnant women
* breast-feeding women
* people under justice protection.

Min Age: 16 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Female patients with anorexia nervosa or bulimia nervosa in many studies and with alexithymia wich is a characteristic found in this patient.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Alexithymia rate using de Toronto Alexithymia Scale | 3 months
  Alexithymia rate using de Toronto Alexithymia Scale (TSA) in 20 items at 3 months. TAS-20 is a self-questionnaire of 20 items rated from 1 (complete disagreement) to 5 (full agreement) evaluating three central dimensions of alexithymia: the difficulty of identifying Difficulties Identifying Feelings (DIF), Difficulties Describing Feelings (DDF), and Externally Oriented, Concrete Thinking (EOT).

SECONDARY OUTCOMES:
Body Mass Index (BMI) evolution for anorexic patient | 3 months
  Body Mass Index (BMI) evolution for anorexic patient at 3 months The lower the Body Mass Index (BMI), the more alexithymia is important. The weight is collected weekly (twice a week at the CHU) the same day in a standardized way: in the presence of a nurse, in the morning on an empty stomach, after going to the bathroom, underwear, and using the same scale . The size is measured in similar conditions with the same meter at the entrance. The BMI is calculated by performing the operation weight divided by height squared and is expressed in kg / m2.
Effect of depression on alexithymia using the Beck Depression Inventory-II | 3 month
  Effect of depression on alexithymia at 3 month, using the Beck Depression Inventory-II (BDI-II) The revised version of the BDI or BDI-II, is a 21-item Likert scale-type self-questionnaire assessing depressive symptoms. These different items are rated from "rarely" (0) to often (3). The total score can be used to rate the severity of depression: 0 to 13 (minimum); 14 to 19 (light); 20 to 28 (moderate); > 28 (severe [78]). Note that there is no validated threshold in adults to define a depressive episode characterized.
  It has a very good level of internal consistency and reproducibility: the Cronbach Alpha coefficient is high from 0.83 to 0.96 according to the studies in a review of the 2013 literature, this is also the case in French
Effect of anxiety on alexithymia using the State Trait Anxiety Inventory-YA | 3 months
  Effect of anxiety on alexithymia at 3 month, using the State Trait Anxiety Inventory-YA (STAI-YA) The STAI is a Likert type self-questionnaire assessing anxiety that includes two scales: the STAI forms Y-A for "anxiety-state" (AE) and the YB form for "anxiety-trait" (AT) . Each scale is composed of 20 propositions: the scale E (State) relative to what the subject feels on the moment and the scale T (Line) relating to what the subject generally feels [81].
  Each item has a score ranging from 1 to 4 (4 being the highest degree of anxiety). We thus obtain the score AE which is the sum of the 20 questions of the page relative to the state and which varies from 20 to 80 as well as the score AT is the sum of the 20 questions of the page "Trait" which also varies from 20 to 80. We will therefore find a very high score (> to 65), high (from 56 to 65), average (from 46 to 55), low (from 36 to 45) or very low (≤35).

CONTACTS AND LOCATIONS:
Overall Officials: Clara Letamendia, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No